CLINICAL TRIAL: NCT02948348
Title: A Phase 1b/2 Multicenter Study to Investigate the Safety, Efficacy and Proof of Concept (POC) of Nivolumab Monotherapy as a Sequential Therapy Following Preoperative Chemoradiotherapy Patients With Locally Advanced Resectable Rectal Cancer
Brief Title: Study to Nivolumab Following Preoperative Chemoradiotherapy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Takayuki Yoshino (Other)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor-Investigator, Takayuki Yoshino, Director of Gastrointestinal Oncology Division, National Cancer Center Hospital East
Organization: National Cancer Center Hospital East (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPOC1504
Record Dates: First submitted 2016-09-08; First posted 2016-10-28 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Cancer of Rectum
MeSH Terms: conditions — Rectal Neoplasms | interventions — Nivolumab; Chemoradiotherapy; Capecitabine; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nivolumab & Ipilimumab(Only Cohort D) (Experimental): chemoradiotherapy with capecitabine+ Nivolumab + Ipilimumab(Only Cohort D) + surgical therapy
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Capecitabine:Dose of 1650mg/m2,14days, Radiation:45Gy/25 fractions, Nivolumab :240mg on day1 of each cycle, Surgical therapy:The resection (LAR), intersphincteric resection (ISR), or abdominoperineal resection (APR).
  Other Names: Opdivo; Chemoradiotherapy with capecitabine; Surgical therapy
Drug: Ipilimumab — For only Cohort D,1 mg/kg at six-week intervals
  Other Names: Yervoy

SUMMARY:
This is a phase Ib/II, open-label, single-arm, multicenter study to investigate the safety, efficacy, and proof of concept (POC) of monotherapy with nivolumab, an anti-PD-1 antibody drug, as a sequential therapy following chemoradiotherapy (CRT) with capecitabine and subsequent surgical therapy in patients with locally advanced resectable rectal cancer.

DETAILED DESCRIPTION:
[Phase Ib]

After preoperative CRT, to sequentially administer nivolumab in combination for patients with locally advanced resectable rectal cancer. To evaluate the safety of nivolumab in sequential combination therapy, the onset of dose-limiting toxicity (DLT) and the safety of subsequent surgical therapy, and to decide on a recommended dose (RD) for the phase II part.

[Phase II] PhaseⅡ is composed of 4 cohorts.

Cohort A: First-onset rectal cancer cohort (42 cases) To evaluate the efficacy and safety of nivolumab (at the RD determined in Phase Ib) in sequential combination with surgery, administered following preoperative CRT.

And to search for biomarkers related to therapeutic effects in first-onset cases. Evaluate the safety of surgical treatment.

Cohort B: Rectal cancer with localized recurrence cohort (10 cases) To conduct an exploratory evaluation of the efficacy and safety of nivolumab (at the RD determined in Phase Ib) in sequential combination with surgery, administered after preoperative CRT.

Search for biomarkers related to therapeutic effects in localized recurrence cases. Conduct an exploratory evaluation on the safety of surgical treatment.

Cohort C: Rectal cancer with resectable lung/liver metastasis cohort (10 cases) To conduct an exploratory evaluation of the efficacy and safety of nivolumab (at the RD determined in Phase Ib) in sequential combination with surgery, administered after preoperative CRT.

Search for biomarkers related to therapeutic effects in resectable lung/liver metastasis cases. Conduct an exploratory evaluation on the safety of surgical treatment.

Cohort D: First-onset rectal cancer using ipilimumab-nivolumab combination cohort (25 cases) To conduct an exploratory evaluation of the efficacy and safety of nivolumab (240 mg/body at two-week intervals) and ipilimumab (1 mg/kg at six-week intervals) after preoperative CRT, and search for biomarkers related to therapeutic effects in first-onset cases. Conduct an exploratory evaluation on the safety of surgical treatment.

ELIGIBILITY:
Inclusion criteria:

(A. Phase Ib and Cohorts A and D only)

A1. Rectal cancer patients who have not undergone treatment for pre-CRT tumors situated 12 cm or less from the lower edge of the AV.

A2. The primary rectal lesion is histopathologically diagnosed as adenocarcinoma.

A3. Pre-CRT clinical stage is clinical T3-4 N-any M0.

A4. Macroscopic radical resection is deemed possible on pre-CRT image diagnosis.

A5. Aged between 20 and 80 years at the time of enrollment.

(B. Cohort B only)

B1. Clinically diagnosed with local recurrence after rectal surgery.

B2. The main site of recurrence is limited to the pelvis by pre-CRT imaging diagnosis.

B3. Macroscopic radical resection is deemed possible on pre-CRT imaging diagnosis.

B4. Aged between 20 and 75 years at the time of enrollment.

(C. Cohort C only)

C1. Rectal cancer patients who have not undergone pretreatment for a pre-CRT tumor which is 12 cm or less from the lower AV.

C2. The primary rectal lesion is histopathologically diagnosed as adenocarcinoma.

C3. The pre-CRT clinical stage is clinical T3-4 N-any M1a (liver) M1a (lungs).

C4. Macroscopic curative resection of the primary rectal lesion is deemed possible on pre-CRT imaging diagnosis.

C5. A metastatic liver tumor or a metastatic lung tumor has been diagnosed as clinically resectable prior to CRT and during clinical trial enrollment.

(D. Common to all cohorts in Phase Ib and Phase II)

D1. Patients who have provided consent through a consent form.

D2. Patients whose Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) is 0 or 1 at the time of enrollment.

D3. CRT was administered:

D4. Patients whose CRT adverse events have recovered to Grade 1 or lower based on CTCAE ver.4.0. within 14 days after the end of CRT, and are expected to be able to take nivolumab (patient is still eligible even if adverse events are not restored to Grade 1, provided that the blood cell count satisfies the eligibility criteria specified in point D8).

D5. Patients with no remote metastases as confirmed by imaging at the end of CRT (testing is allowed from 14 days before the end of CRT to the trial enrollment date).

D6. For women who may become pregnant (including patients who are not menstruating due to chemically-induced menopause among other medical reasons), patients who agree to use contraception for at least 23 weeks after the last administration of the investigational drug, starting from the day they provide consent (30 days (ovulation cycle) plus five times the elimination half-life of the investigational drug).

D7. For men, patients who agree to use contraception for at least 31 weeks after the last administration of the investigational drug, starting from the day they provide consent (90 days (spermatogenesis cycle) plus five times the elimination half-life of the investigational drug).

D8. Patients who have the sufficient organ function at the time of enrollment.

Exclusion criteria

1. Patients diagnosed with active double cancer (synchronous double cancer and double cancer with disease-free period within five years from enrollment).

   However, lesions equivalent to intraepithelial or mucosal carcinoma deemed cured by localized treatment are not classified as active double cancer.
2. Patients with a history of pelvic irradiation prior to this rectal cancer treatment.
3. Patients who have not given consent through the informed consent form.
4. Patients deemed by the investigator to be ineligible for the trial.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-10; Primary Completion 2021-12 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | 1 year
  Pathological complete response will be evaluated with American Joint Committee on Cancer (AJCC) Cancer Staging

SECONDARY OUTCOMES:
Objective response rate | 1 year
  Evaluation Criteria In Solid Tumors (RECIST)
Recurrence pattern (local or distant) | 1 year
Disease-free survival (DFS) | 5years
  Evaluation Criteria In Solid Tumors (RECIST)
Overall survival (OS) | 5years
  Evaluation Criteria In Solid Tumors (RECIST)
Incidence of adverse events (AEs) | 1 year
  Safety will be evaluated with CTCAE v4.0
Rate of completing the protocol therapy | 1 year
Rate of radical resection | 1 year
Safety evaluation | 5years
  Safety will be evaluated with CTCAE v4.0
macroscopic evaluation of (rectal cancer) resected specimen | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Takayuki Yoshino, Dr, Study Chair — Gastrointestinal Oncology Division National Cancer Center Hospital East
Locations (3):
- Japan (3):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Hokkaido University, Sapporo, Hokkaido
  - Osaka National Hospital, Osaka

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tsukada Y, Bando H, Inamori K, Wakabayashi M, Togashi Y, Koyama S, Kotani D, Yuki S, Komatsu Y, Homma S, Taketomi A, Uemura M, Kato T, Fukui M, Nakamura N, Kojima M, Kawachi H, Kirsch R, Yoshida T, Sato A, Nishikawa H, Ito M, Yoshino T. Three-year outcomes of preoperative chemoradiotherapy plus nivolumab in microsatellite stable and microsatellite instability-high locally advanced rectal cancer. Br J Cancer. 2024 Jul;131(2):283-289. doi: 10.1038/s41416-024-02730-7. Epub 2024 Jun 4. PMID 38834744